CLINICAL TRIAL: NCT03434899
Title: Effects of Physical Activity With Online Support for Individuals With Chronic Widespread Pain (CWP)
Acronym: GAU-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOU VGR 237261
Record Dates: First submitted 2018-02-06; First posted 2018-02-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Widespread Pain
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Health care plan including physical exercise and online support during the entire study
  Interventions: Behavioral: Physical exercise and online support
- Control Group (Active Comparator): Health care plan including physical exercise
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise and online support — Person-centered design of a health care plan including individually adjusted physical exercise. Online support for management of health care plan.
  Arms: Intervention group
Behavioral: Physical exercise — Person-centered design of health care plan individually adjusted physical exercise.
  Arms: Control Group

SUMMARY:
The aim is to evaluate a novel treatment routine where contact through a smart phone/computer is used for online support for patients suffering from chronic widespread pain (CWP). The outline is that patients are encouraged to perform physical activity during a period of 12 months with online support from a physical therapist.

DETAILED DESCRIPTION:
The intervention follows principles from the theories of person-centered care and self-efficacy. The examinations performed at baseline and after six months were conducted by blinded examiners at a visit at the primary health care centers. All participants developed a person-centered health plan for physical activity together with a physiotherapist. The intervention group was supported with a digital platform for six months.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the American Colleague of Rheumatology (ACR) 1990 criteria for chronic widespread pain (CWP)
* access to a smart phone or computer

Exclusion Criteria:

* other serious diseases that cause pain or hinder exercise, such as heart disease, neurological disease or severe osteoarthritis
* unable to speak or read Swedish

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Pain during the last week | Change from Baseline Pain at 6 months
  The Fibromyalgia Impact Questionnaire (FIQ) subscale for pain.

SECONDARY OUTCOMES:
Fatigue | Change from Baseline Fatigue at 6 months
  The Multidimensional Fatigue Inventory (MFI-20), comprising several subscale, of which the Physical Fatigue subscale is of interest for this study.
Health | Change from Baseline Health at 6 months
  The Fibromyalgia Impact Questionnaire (FIQ) total score. The FIQ comprises 10 subscales and the total score is the mean value of them.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Mannerkorpi, PhD, Principal Investigator — Sahlgren University Hospital
Locations (3):
- Sweden (3):
  - Alingsas Primary Health Care, Alingsås
  - Göteborg Primary Health Care, Gothenburg
  - Uddevalla Primary Health Care, Uddevalla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldthusen C, Bergenheim A, Barenfeld E, Gjertsson I, Larsson A, Mannerkorpi K. Experience of co-creation of a health plan and support for sustainable physical activity among people with chronic widespread pain: a qualitative interview study in Sweden. BMJ Open. 2022 Apr 8;12(4):e059432. doi: 10.1136/bmjopen-2021-059432. PMID 35396312